CLINICAL TRIAL: NCT02602561
Title: Effects of HMB Supplementation on Muscle Mass Following ACL Reconstructive Surgery
Brief Title: Effects of HMB Supplementation on Recovery Following ACL Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metabolic Technologies Inc. (Industry)
Collaborators: Iowa State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MTI2015-CS02
Record Dates: First submitted 2015-11-06; First posted 2015-11-11 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: ACL Injury
Keywords: HMB; beta-hydroxy-beta-methylbutyrate; ACL; surgery; muscle mass
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — beta-hydroxyisovaleric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HMB (Active Comparator): 3 g HMB/day
  Interventions: Dietary Supplement: HMB
- Placebo (Placebo Comparator): Placebo administered similar to the active comparator
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: HMB
  Other Names: beta-hydroxy-beta-methylbutyrate
  Arms: HMB
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The anterior cruciate ligament (ACL) is a primary stabilizer of the knee, and thus when ACL injury occurs participation in physical activity is compromised. Reconstructive surgery is often necessary to repair the damage which is then followed by a regimen of physical therapy in order to regain full activity. Nutritional intervention after the surgery could help the patient maintain muscle mass during recovery, thus allowing for a quicker return to normal activity.

DETAILED DESCRIPTION:
Beta-hydroxy-beta-methylbutyrate (HMB) is a nutritional supplement shown to improve muscle mass with exercise, and also in muscle loss conditions caused by a decrease in physical activity. Participants will be recruited who will undergo reconstructive surgery for a complete ACL tear and will then enter a standard physical therapy program during a six week recovery period. Subjects will receive either HMB or a placebo supplement during the recovery period. Muscle mass will be measured two weeks prior to the surgery and again after the recovery period using an InBody 720 body composition analyzer. Additionally, the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire will be administered as a measure of recovery and activity level during the study.

ELIGIBILITY:
Inclusion Criteria:

* Complete anterior cruciate ligament (ACL) tear
* Will benefit from ACL reconstructive surgery
* Are able to participate in the physical therapy program
* No previous major knee injuries or surgeries
* No health conditions affecting muscle mass

Exclusion Criteria:

* Incomplete ACL tear
* Have multiple or bilateral ligament tears
* Are unable to participate in the physical therapy program
* Have had previous major knee injuries or surgeries
* Have health conditions affecting muscle mass

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2015-11; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Skeletal Muscle Mass by impedance measurement using the InBody 720 body composition analyzer | Six Weeks
  Measurement of muscle mass will indicate if the active comparator has preserved or increased muscle mass during the post-surgical recovery period.

CONTACTS AND LOCATIONS:
Overall Officials: John A Rathmacher, PhD, Principal Investigator — Metabolic Technologies Inc.
Locations (1):
- Iowa State University, Ames, Iowa, United States